CLINICAL TRIAL: NCT02548481
Title: Validation and Standardisation of a Pool of Simplified Evaluation Aimed to the Diagnoses of Aphasic Disorders and Adapted to the Patients Suffering an Acute Phase of Stroke
Acronym: BESTA-AVC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: I14004
Record Dates: First submitted 2015-09-09; First posted 2015-09-14 (Estimated); Last update posted 2020-06-01 (Actual); Status verified 2020-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- BESTA scale: BESTA scale is administered at T0, T1 (3 months) and T2 (1 year)
  Interventions: Other: BESTA scale

INTERVENTIONS:
Other: BESTA scale — BESTA scale is administrated at T0, T1 and T2.

SUMMARY:
Every year in France, from 100 000 to 145 000 people are affected by a stroke. 75% patients survived with aftereffects, in particular aphasic disorders.

A sketch of a new tool called BESTA aiming to a rapid handover to the acute phase post stroke had been worked out. After a meeting, 13 multidisciplinary experts have discussed, adjusted and a new complete tool (BESTA) had been created in order to evaluate the different states of aphasia.

The goal of this study is the validation and the standardization of this new BESTA tool.

ELIGIBILITY:
Inclusion Criteria:

Patients with stroke:

* Every patient over 18,
* admitted among neuro-vascular unit,
* native french speaker,
* the level of vigilance is satisfactory in order to allow a speech therapy test.

Healthy Volunteers:

* Every volunteers over 18,
* without any medical history of a stroke or any speech disorders,
* native french speaker.

Exclusion Criteria:

Patients with stroke and Healthy Volunteers :

* dementia disease
* psychiatric condition
* non-equipped deafness
* pregnant woman
* patient with medical histories of stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Administration of BESTA scale (test to assess) within 3 days after stroke and at 3 months and 1 year after stroke. This scale will be compared to standard scales.
Sampling Method: Probability Sample
Enrollment: 395 (Estimated)
Dates: Start 2015-11; Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
validity of concomitant criterion at T0 versus LAST | 1 day
  T0: the gold standard was determined by the expert group is the LAST screening tool.
  The tool to be evaluated is the BESTA at T0. However, as written expression is not evaluated in the LAST, only the dimensions and Oral Expression Listening Comprehension of BESTA may actually be faced with LAST scale.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco MACIAN, MD, Principal Investigator — University Hospital, Limoges
Locations (1):
- Limoges Hospital, Limoges, France